CLINICAL TRIAL: NCT04024293
Title: A Prospective Single Center Open Label Study Assessing Intraocular Pressure Measurements Using a Novel Sensing Contact Lens-based Device as Compared to Standard Tonometry, in Open Angle Glaucoma and Ocular Hypertensive Patients
Brief Title: Intraocular Pressure Measured by a Novel Sensing Contact Lens Versus Tonometry
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sensimed AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GF-1801-S
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All participants (Experimental): All patients will be follow the same procedures and be placed the investigational device
  Interventions: Device: Goldfish (GF)

INTERVENTIONS:
Device: Goldfish (GF) — The GF lens (SCL) will be place on participant's eye for a 24h IOP recording session

SUMMARY:
While elevated intraocular pressure (IOP) is no longer part of the definition of glaucoma it remains the sole proven modifiable risk factor for the onset and progression of glaucoma.

IOP is known to vary with the time of day as well as with daily activities. The importance of the nycthemeral IOP pattern for successful management of glaucoma has been well documented, especially for patients who experience visual loss despite apparently normal and/or controlled IOP during office hours.

The current way of assessing nycthemeral IOP fluctuation is to perform repeated discrete tonometry measurements, once per hour in the best cases. Since its development in the 50s, Goldmann applanation tonometry (GAT) has remained the gold standard method for measuring IOP, despite its limitations. However, tonometry may be an imperfect method for measuring changes in IOP because it allows only snapshot and non-continuous measurements, it is not physiologic and disturbs the sleep architecture.

There have been many efforts in the past decades to search for an ambulatory and frequent method to monitor IOP for 24 hours. In this context, Sensimed AG has recently developed a sensing contact lens-based device intended to measure IOP over 24 hours, the Goldfish (GF).

First-in-man data obtained with this device showed agreements between IOP measured by GF and values obtained by standard tonometry in the same eye, comparable to literature results for routinely used tonometry devices. However, this pilot study included 9 subjects only with improvable safety, tolerability and efficacy profiles.

The main goal of this study is to assess IOP measurements with the GF and compare the values with those obtained by standard tonometry in patients with open angle glaucoma (OAG) and ocular hypertension (OHT).

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* A clinical diagnosis of primary open angle glaucoma (POAG), including normal tension glaucoma (NTG), for OAG patients
* A clinical diagnosis of OHT, for OHT patients
* For all patients:

Open angles on gonioscopy Aged ≥ 18 years, either gender Both central corneal radii (CCR) between 7.3mm (46.23D) and 8.05mm (41.93D), with a maximum difference of 2D between the 2 radii in the study eye Central corneal thickness (CCT) between 490µm and 600µm in the study eye

Exclusion Criteria:

* Ocular pathology (other than glaucoma or OHT)
* Previous glaucoma, cataract or refractive laser/surgery
* Corneal or conjunctival abnormality, precluding contact lens adaptation
* Insufficiency of lacrimal secretion
* Subjects with allergy to corneal anesthetic
* Subjects with contraindications for silicone contact lens wear
* Subjects with contraindications for Diamox or Latanoprost or Timolol
* Skin irritations, skin eczema or other indications against the wearing of adhesive patches
* Subjects unable or unwilling to comply with the study procedures
* Subjects lacking the capacity to consent (vulnerable persons)
* Subjects with history of cardiac failure, treated cardiopathy or renal failure
* Subjects with known cognitive disorders
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
GF IOP measurement as compared to IOP | 24 hours
  Differences between GF IOP measurements at the recording start/end and the values obtained by GAT before/after GF SCL placement/removal, in the same eye

CONTACTS AND LOCATIONS:
Overall Officials: Kaweh Mansouri, Pr, Principal Investigator — Swiss Glaucoma Foundation
Locations (1):
- Clinique Montchoisi, Lausanne, Canton of Vaud, Switzerland